CLINICAL TRIAL: NCT03126747
Title: Drug Use Investigation (DUI) of YazFlex for Endometriosis-associated Pelvic Pain and/or Dysmenorrhea
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18703
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis and Dysmenorrhea
MeSH Terms: conditions — Endometriosis; Dysmenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAY86-5300_YAZ-Flex: Patients with endometriosis-associated pelvic pain or dysmenorrhea
  Interventions: Drug: BAY86-5300_YAZ-Flex

INTERVENTIONS:
Drug: BAY86-5300_YAZ-Flex — Patients with endometriosis-associated pelvic pain and/or dysmenorrhea are enrolled solely after the physician's decision of YazFlex treatment in routine clinical practice.

SUMMARY:
This study is a Japanese post-marketing surveillance (PMS) which is required by the regulatory authorities. General objective of PMS is to confirm the clinical usefulness, especially the safety profile of a drug under the routine clinical practice.

DETAILED DESCRIPTION:
It is a local, non-interventional, multi-center, single-cohort study using primary data of patients treated with YazFlex in endometriosis or dysmenorrhea indication.

A total of 600 patients (300 for endometriosis and 300 for dysmenorrhea) is planned to be enrolled in 2 years.

The treatment should be performed in Japan based on the product label. The patients will be observed for up to 2 years (1 year at the earliest) during their YazFlex treatment.

The outcome variables for the primary objective are treatment emergent adverse events (TEAEs) and adverse drug reactions (ADRs). The outcome variables for the secondary objective include newly developed haemorrhagic ovarian cyst, genital bleeding, severity of dysmenorrhea, pelvic pain and compliance status in the new flexible regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endometriosis-associated pelvic pain and/or dysmenorrhea.
* Patients for whom the decision to initiate treatment with YazFlex is made as per physician's clinical practice.

Exclusion Criteria:

- Patients participating in an investigational program with interventions outside of routine clinical practice.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Endometriosis-associated pelvic pain and/or Dysmenorrhea
Sampling Method: Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reactions (ADRs) | Up to 2 years ( 1 year at the earliest)
  Events will be summarized by frequency tables (e.g. absolute and relative frequencies) using the MedDRA cording system.

SECONDARY OUTCOMES:
Incidence proportions of YAZ-Flex therapy | Up to 2 years ( 1 year at the earliest)
Incidence proportions of extent of bleeding | Up to 2 years ( 1 year at the earliest)
Incidence proportions of treatment suspension | Up to 2 years ( 1 year at the earliest)
  The duration of suspension is defined as a period of at least 3 consecutive days of treatment suspension.
Number of days with menstrual pain | Up to 2 years ( 1 year at the earliest)
  Menstrual pain is continuous menstrual pain or lower abdominal pain that is observed for menstruation or withdrawal blood events and may spread to the back or thigh. Pain may be recognized 2 days before bleeding, and ends by the last day of menstruation or withdrawal.
Number of date of using analgesic | Up to 2 years ( 1 year at the earliest)
  Record the date of using the analgesic.
Change in severity of dysmenorrhea | Up to 2 years ( 1 year at the earliest)
  The severity will be evaluated and recorded the following criteria.
  1. None
  2. Somewhat obstructing work (school or housework)
  3. get a problem with one's work (studies / housework) because the more one wants to lie down
  4. Fall asleep for more than 1 day, and cannot do one's work (school or housework)
Change in severity of pelvic pain by using Numeric Rating Scale (NRS) | Up to 2 years ( 1 year at the earliest)
  The degree of pelvic pain in each menstrual period, menstrual period, sexual intercourse and defecation will be evaluated using NRS score (11 levels from no pain is "0" to highest pain "10" ) in each month.
Change in quality of Life by using EQ-5D-5L , EIS and/or MDQ | Up to 2 years ( 1 year at the earliest)
  Endometriosis Impact Scale (EIS) (for disease burden of endometriosis) Menstrual Distress Questionnaire (MDQ) (for disease burden of dysmenorrhea) EQ-5D (for general QOL measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Yoshino O, Suzukamo Y, Yoshihara K, Takahashi N. Quality of Life in Japanese Patients with Dysmenorrhea or Endometriosis-Associated Pelvic Pain Treated with Extended Regimen Ethinylestradiol/Drospirenone in a Real-World Setting: A Prospective Observational Study. Adv Ther. 2022 Nov;39(11):5087-5104. doi: 10.1007/s12325-022-02301-3. Epub 2022 Sep 2. PMID 36053449
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/